CLINICAL TRIAL: NCT01898195
Title: Improving Adherence to Smoking Cessation Medication Among PLWHA
Acronym: HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-02165
Record Dates: First submitted 2013-07-01; First posted 2013-07-12 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (Active Comparator): Participants in this arm will receive varenicline for smoking cessation.
  Interventions: Drug: Varenicline
- Standard Care + Text message (Experimental): Participants in this arm will receive varenicline, plus twice daily adherence/motivational texts.
  Interventions: Drug: Varenicline; Behavioral: Text Message
- Standard Care + Text Message + ABT (Experimental): Participants in this arm will receive varenicline, plus twice daily adherence/motivational texts and seven phone developed Adherence Behavioral Therapy sessions
  Interventions: Drug: Varenicline; Behavioral: Text Message; Behavioral: Adherence Behavioral Therapy

INTERVENTIONS:
Drug: Varenicline — Varenicline will be provided for three months.
  Other Names: Chantix
Behavioral: Text Message — Text messages will be developed twice daily for three months
  Arms: Standard Care + Text Message + ABT; Standard Care + Text message
Behavioral: Adherence Behavioral Therapy — Seven Adherence Behavioral Therapy sessions will given over a three month period
  Other Names: ABT
  Arms: Standard Care + Text Message + ABT

SUMMARY:
Smoking rates among individuals living with HIV/AIDS range between 47% and 65%, a prevalence that is roughly three times the rate of the general population. This elevated prevalence is alarming given the increased likelihood of numerous adverse health outcomes experienced by HIV-positive smokers. Cigarette smoking is associated with greater levels of HIV-related symptom burden and appears to decrease the effectiveness of HAART as assessed by both viral load and CD4 counts (Vidrine 2009, Marshall 2009, Vidrine 2007, Miguez-Burbane 2005). PLWHA who smoke are also at increased risk of infections and noninfectious pulmonary complications and both AIDS-associated and non-AIDS-associated malignancies compared to nonsmokers. This study will refine and pilot test a theory-driven smoking cessation intervention that enhances existing behavioral approaches by testing the impact of text message reminders to take varenicline and the feasibility and additional impact of including adherence-focused behavioral cessation counseling. The investigators propose to randomize 190 participants, recruited from three HIV/AIDS clinic, to a three arm pilot study that compares: 1) Standard Care (SC), 2) SC + text message reminders, and 3) SC + text message reminders + cell phone-delivered adherence-focused behavioral therapy (ABT). Participants in all three arms will receive varenicline for 12 weeks. The primary outcomes are adherence to varenicline and biochemically validated smoking abstinence at 12 weeks and 3-month follow-up from the time of study enrollment.

DETAILED DESCRIPTION:
To accomplish the study's aims the investigators propose a three phase study: PHASE 1) Formative phase (n=40) to pretest text messages and to explore barriers to cessation and adherence to cessation medication; PHASE 2) a Pretest phase (n=10) to test and revise the intervention components and to assess design issues that may emerge, including those associated with contacting subjects via cell phone, participant capacity to view text messages, timing and content of text messaging, and use of the eCAPs system; and PHASE 3) a Pilot randomized control trial (RCT) in which the investigators will randomize 190 participants, recruited at St. Luke's Roosevelt Comprehensive Care Clinics, to a three-arm study that compares: 1) Standard care (SC), which includes receiving varenicline and brief counseling; 2) SC + daily text messages medication reminders (TxT); or 3) SC + TxT + seven sessions of cell-phone-delivered, adherence-focused behavioral therapy (ABT). Text messages will include medication reminders and motivational messages related to adherence and maintaining abstinence. Participants in all three arms will receive varenicline for 12 weeks. To have a total sample of 150 subjects through the end of treatment at 12 weeks, or 50 subjects in each arm, the investigators will randomize 190 patients to account for a 20% attrition rate. Subjects will be surveyed at six time points including the baseline assessment.

PHASE 1: FORMATIVE EVALUATION Focus groups with patients. Focus groups (lasting from 60 to 90 minutes) will be conducted with HIV+ smokers. To recruit patients for Phase 1, research assistants will approach all individuals within the clinic setting to screen for tobacco use. If they are a current smoker they will be asked if they wish to participate in a scheduled focus group at a convenient time. The research assistants will recruit 80 patients and expect to complete 4 focus groups with 10 participants in each for a total of 40 participants. The main aims of these focus groups are: 1) to obtain feedback on the text message library to determine which messages will be most acceptable and useful, and how often the patients would like to receive messages; 2) to assess comfort with using the pre-paid phone to receive and send messages; 3) to assess confidentiality concerns regarding receiving the text messages and how the patients may be edited to avoid loss of confidentiality; and 4) to explore attitudes and beliefs about varenicline, previous experiences using varenicline, potential challenges with adhering to varenicline, and similarly to explore experiences with past quit attempts and barriers (individual, social, structural) to quitting.

The focus groups will follow written guides. In addition to pre-specified domains drawn from the research questions above, the group facilitator will also listen for and explore emergent topics. Focus groups will be audio-recorded and two research assistants will take notes during each group discussion. All audio recordings will be transcribed verbatim, and transcripts will be supplemented with notes taken during the focus group to ensure accuracy. These transcripts will be analyzed for both pre-determined and emergent themes.

PHASE 2: PRE TEST Prior to starting the RCT the investigators will pre-test the intervention components (ARM 3) to assess study design issues that may emerge, including those associated with contacting subjects via cell phone, participant capacity to view text messages, timing and content of text messaging, and use of the eCAPs system. Ten patients will be enrolled for this phase with a target sample of 6 at end-of-treatment. Quantitative data collection, described below, will follow. The investigators will also conduct post-intervention in-depth interviews with all enrolled subjects to obtain feedback on the components' utility, acceptability, and safety. The research team and consultants will meet after this pilot test to make adjustments to the intervention components prior to the RCT.

PHASE 3: PILOT RCT Overview. This phase of research will compare three smoking cessation interventions that were tested and refined in Phases 1 and 2. A total of 190 PLWHA who are patients at CCC will be screened for this phase with a target sample of 150 at end-of-treatment. The investigators will use a randomized controlled trial design. This is not a formal efficacy trial but a test of the interventions feasibility, safety, and acceptability. Additionally the study will provide preliminary evidence of efficacy of the intervention components with respect to the study's main endpoints: a) adherence to varenicline and b) smoking abstinence at 12 and 24 weeks. This data will inform the design of a larger R01.

Intervention conditions ARM 1: Standard Care (SC). All CCC patients are screened for tobacco use during their routine visits and offered a referral to the New York State (NYS) Quitline. As part of current standard care, all trial participants will receive a self-help information sheet, tailored to HIV+ smokers with frequently asked questions about using varenicline, and a wallet card with the State Quitline number. All subjects will be offered varenicline for 12 weeks. All study participants will be asked whether they prefer to receive phone calls and text messages from the study staff via their own phone or a phone provided by the study, at no cost to the participant. If they choose the latter option, they will be given a pre-paid cell phone for 3 months. Subjects in the SC arm will receive phones to facilitate their ability to call the Quitline for assistance and to enable us to send follow-up appointment reminders via text message. Each pre-paid phone will have an allowance of 200 minutes and unlimited text messages per month. The investigators will instruct participants to use their minutes only toward tobacco treatment or study related purposes. The investigators will track minutes used and if minutes are used out, the investigators will add just enough minutes when they need to contact the subject.

Varenicline therapy: All patients enrolled in the study will be given a 12-week supply of varenicline. The dose will be 0.5 mg/day for 3 days followed by 0.5 mg BID for the next 4 days, and 1 mg BID after first 7 days. The research assistant will explain the use of the medication, review potential side effects, and provide each subject with a wallet size instruction card that will have the dosing schedule and information on how to use the medication. Subjects will receive the medication at a follow-up study visit one week after they are consented. Subjects will receive a three-week supply of varenicline and return at week 4 of the study (timed from the first week they receive the medication). At the week 4 visit they will receive another 4 weeks of medication and will be asked to return at week 8 to receive the final 4 weeks of medication. More than one eCAP bottle will be distributed, depending on the dose of medication and the week of treatment.

ARM 2: SC + Text messages (TxT). Subjects randomized to this arm will receive SC plus twice daily text messaging to remind them to take their medication. Participants will begin receiving text messages the day before they start taking medication, and text messaging will continue for 12 weeks. The text messages are designed to convey relevant information to the subjects while permitting a protective ambiguity. For example, none of the messages transmitted to participants will use the terms HIV or AIDS. In addition, each text message will have the tag "ACT" (Adherence to Cessation Treatment) indicating that it is coming from the study. Participants will receive one medication adherence reminder message and one motivational message regarding tobacco cessation each day. RTI staff will monitor the delivery of the text messages. If participants do not receive text messages for two consecutive days, the study research assistant will call them to assess reasons for message failure. During the study, participants may opt out of receiving any category of messages by contacting the study research assistants and informing him/her of their request. Requests to decline a specific message type or to fully withdraw from the study will be handled promptly and subjects will stop receiving messages within 48 hours of submitting their request to the study research assistant. The investigators will use both symbols and text to accommodate low literacy levels.

ARM 3: SC + TxT + adherence-focused motivational and behavioral therapy (ABT). In addition to SC and TxT, the behavioral intervention group will receive seven proactive cell-phone-delivered counseling sessions over a 6-week period. Drs. Shelley and Krebs have adapted the telephone counseling manual that was developed and tested by Dr. Sherman which was based on Dr. David Kalman's "Treatment Manual for Extended Counseling to Treat Tobacco Addiction,". The draft manual will be reviewed by Drs. Sherman, Wolfe, and Morgenstern and then revised prior to the Phase 2 pretest. The research team will meet again to further revise the manual based on findings from the Phase 2 post-intervention qualitative interviews. The content of the manual combines the principles of Cognitive Behavioral Therapy (CBT) with Motivational Interviewing (MI) techniques, both of which have been applied to smoking cessation with promising results.

ELIGIBILITY:
Inclusion Criteria:

1. Current patient at one of two SLR CCC clinics with a designated physician (had intake visit and enrolled into clinic)
2. Age 18 years or older;
3. Current or regular smoker (>5 cigarettes per day);
4. Carbon Monoxide (CO) monitor reading of >8 ppm;
5. Willingness to set a quit date;
6. Able to conduct activities in English;
7. Ability to provide informed consent;
8. Willingness to carry/use a cell phone; AND
9. Eligible to take varenicline as determined by the patient's primary care provider

Exclusion Criteria:

1. Unstable cardiovascular disease (e.g. uncontrolled blood pressure, unstable angina, or myocardial infarction in the past 4 weeks);
2. Current homicidal or suicidal ideation, history of suicidal ideation, or history of psychosis;
3. Has a serious or untreated psychiatric illness (major depression, bipolar or schizophrenia);
4. Severe renal impairment (defined as having a creatinine clearance < 30mL/min);
5. Currently using smokeless tobacco;
6. Currently using FDA-approved smoking cessation medication or other smoking cessation treatment and or participating in another smoking cessation program;
7. Active drug use identified by a score of 6 or above on DAST-10 Drug Abuse Screening Test;
8. Alcohol dependence or risk drinking identified by a score of 5 or above for men and 4 or above for women on AUDIT-C Alcohol Use Disorders Identification Test
9. Pregnant or nursing; AND/OR
10. Has a cognitive impairment that would preclude giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD MPH, Principal Investigator — NYU School of Medicine
Locations (1):
- Spencer Cox Center for Health, New York, New York, United States

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Shelley D, Tseng TY, Gonzalez M, Krebs P, Wong S, Furberg R, Sherman S, Schoenthaler A, Urbina A, Cleland CM. Correlates of Adherence to Varenicline Among HIV+ Smokers. Nicotine Tob Res. 2015 Aug;17(8):968-74. doi: 10.1093/ntr/ntv068. PMID 26180221

RESULTS

PARTICIPANT FLOW:
Period: Varenicline Adherence
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT
Started | 53 | 54 | 51
Completed | 18 | 16 | 15
Not Completed | 35 | 38 | 36
Period: Smoking Abstinence
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT
Started | 53 | 54 | 51
Completed | 18 | 16 | 15
Not Completed | 35 | 38 | 36
Not completed — Did not have good measurements | 35 | 38 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT | Total
Number analyzed (Participants) | 53 | 54 | 51 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 51 | 158
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.64 (10.77) | 46 (9.96) | 47.88 (8.69) | 46.84 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 8 | 32
  Male | 39 | 44 | 43 | 126
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 51 | 158

OUTCOME MEASURES:

1. Primary Outcome: End-of-intervention Varenicline Adherence
Description: number of participants who took at least 80% prescribed dose since last interview, based on pill count
Time Frame: 4 Weeks
Measure: Number; unit: participants
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT
Number analyzed (Participants) | 50 | 53 | 50
participants | 18 | 16 | 15

2. Secondary Outcome: End-of-intervention Smoking Abstinence
Description: number of participants who achieved smoking abstinence based on self-reported 7-day point prevalence smoking abstinence verified by a carbon monoxide (CO) < 8 ppm
Time Frame: 7 Days
Measure: Number; unit: participants
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT
Number analyzed (Participants) | 53 | 54 | 51
participants | 3 | 2 | 8

ADVERSE EVENTS:
Arm/Group | Standard Care | Standard Care + Text Message | Standard Care + Text Message + ABT
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 9/53 | 2/54 | 7/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=53) | Standard Care + Text Message (N=54) | Standard Care + Text Message + ABT (N=51)
Nausea (General disorders) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Changes in appetite (General disorders) | 2 (2) | 0 (0) | 1 (1)
Vivd dreams or nightmares (General disorders) | 2 (2) | 0 (0) | 3 (3)
Problem with sleeping (General disorders) | 3 (3) | 0 (0) | 2 (2)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0) | 0 (0)
Leg Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No